CLINICAL TRIAL: NCT00907972
Title: Effect of Vitamin D3 Supplementation in Parkinson's Disease Patients - A Pilot Study
Brief Title: The Effects of Vitamin D and Bone Loss in Parkinson's Disease
Acronym: PDVD3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Medical Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MMC 08-30
Record Dates: First submitted 2009-05-22; First posted 2009-05-25 (Estimated); Last update posted 2013-07-12 (Estimated); Status verified 2013-07

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; Parkinson Disease; PD; Movement Disorder
MeSH Terms: conditions — Parkinson Disease; Movement Disorders | interventions — Cholecalciferol; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D3 supplementation (Experimental): 1000 IU/day of Vitamin D3
  Interventions: Dietary Supplement: Vitamin D3
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — Vitamin D3
  Other Names: Vitamin D; Vit D; Vit D3
  Arms: Vitamin D3 supplementation
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Health care burdens from neurodegenerative diseases are expected to increase disproportionately. Increasing age also predisposes this same population to other chronic diseases including osteoporosis, a progressive systemic skeletal disease characterized by low bone mass, which leads to an increase susceptibility to fractures. In the United States, 44 million people are estimated to be at risk for osteoporosis and low bone mass emphasizing the enormity of this public health problem.

Parkinson's disease is a progressive neurodegenerative disorder affecting about 1 million people. Evidence indicates that Parkinson's disease patients are at a higher risk for low bone mineral density, which can contribute to increased fractures compared to healthy subjects. In fact, several risk factors of osteoporosis in patients with PD have been identified, including advanced stages of PD, low body mass index, inadequate sunlight exposure and decreased vitamin D levels. Some or all of these factors in conjunction with decreased immobilization that may occur with PD, put patients at increased risks for fractures. Few studies however have examined bone markers in PD patients. Even fewer studies have examined the impact of Vitamin D supplementation on bone metabolism and mineralization in PD patients.

Vitamin D is an essential component in bone health, promoting calcium absorption in the gut and maintaining adequate serum calcium and phosphate concentrations, which enable normal mineralization of bone.

DETAILED DESCRIPTION:
Parkinson's disease is the second most common neurodegenerative disorder after Alzheimer's disease affecting approximately 1% of the population older than 50 years. There is a worldwide increase in disease prevalence due to the increasing age of human populations. The disease is characterized by tremor, stiffness of the limbs and trunk, impaired balance and coordination, and slowing of movements, leading to immobility and frequent falls. Patients also sometimes develop other symptoms, including difficulty swallowing, disturbed sleep, and emotional problems. Parkinson's disease results from the loss of dopaminergic neurons in the substantia nigra region of the brain. The cause and mechanism of continued neuron cell death in the substantia nigra is currently unknown.

Epidemiological studies suggest an association between Parkinson's disease and osteoporosis, vitamin D inadequacy and altered bone and mineral metabolism. Accumulating evidence indicates that patients with Parkinson's disease are at a higher risk for fractures compared to healthy subjects. This could be attributed to several contributing factors including increased rate of falls, vitamin D deficiency, reduced body mass index and reduced bone mineral density.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be >18 yrs of age
* Subject must have a diagnosis of Parkinson's disease (Hoehn and Yahr stages I-III), confirmed by the study physician designated to complete patient staging
* Subject must sign the informed consent documentation according to MMC's IRB guidelines
* Subject must be willing and able to complete all study requirements at the designated time intervals
* Subject must agree to be randomized
* If subject has been taking a separate Vitamin D supplement other than a multivitamin within the last 6 months, the subject must be willing to discontinue Vitamin D supplement for 3 months before entering the study
* Subject must have a vitamin D level greater than 10 ng/mL
* Subjects must have a serum calcium level within the range of 8.4-10 mg/dl.
* Females subjects of child bearing potential must have a negative urine pregnancy test or have undergone a sterilization procedure

Exclusion Criteria:

* Subjects < 18 years old
* Parkinson's disease patients with Hoehn and Yahr stages IV-V.
* Subjects not willing and able to complete all study requirements at the designated time intervals
* Subjects who do not agree to be randomized
* Subjects receiving treatment with bisphosphonates (more that 3 months), parathyroid hormones (PTH) or PTH derivatives, e.g. Teriparatide or Fluoride, in the last 6 months.
* Subjects with an allergy to the investigational product.
* Subjects who have a vitamin D level less than 10 ng/mL
* Subjects who do not have a serum calcium level within the range of 8.4-10 mg/dl.
* Subjects who are pregnant, verified by a urine pregnancy test*

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Direct changes in bone formation and resorption will be investigated by measuring serum 25-hydroxyvitamin D [25(OH)D] level,serum parathyroid hormone (PTH) levels, serum osteocalcin, and serum n-telopeptides (N-Tx) | 12 months

SECONDARY OUTCOMES:
Serum clacium will be measured to monitor for hypercalcemia. | 12 months
Using the Unified Parkinson's Disease Rating Scale (UPDRS) to assess the impact of vitamin D supplementation on PD symptoms | 12 months
Using the Parkinson's Quality of Life measure (PD QoL) to examine the effect of vitamin D supplementation on quality of life | 12 months
Conducting a brief falls assessment to track the incidence of falls throughout the duration of the study | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Plank, MD, Principal Investigator — Conemaugh Health System; Prema Rapuri, PhD, Principal Investigator — Conemaugh Health System
Locations (1):
- Conemaugh Health System - John P Murtha Neuroscience and Pain Institute, Johnstown, Pennsylvania, United States